CLINICAL TRIAL: NCT07177820
Title: Video-Guided Acupuncture Imagery Treatment in Chemotherapy-induced Peripheral Neuropathy
Brief Title: VGAIT for Chemotherapy-induced Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-307
Record Dates: First submitted 2025-07-21; First posted 2025-09-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Intervention Model Description: Video-Guided Acupuncture Imagery Treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VGAIT (Experimental)
  Interventions: Other: Video-Guided Acupuncture Imagery Treatment (VGAIT)

INTERVENTIONS:
Other: Video-Guided Acupuncture Imagery Treatment (VGAIT) — Participants watch a video of acupuncture being applied to the body while simultaneously imagining that it is being administered to them

SUMMARY:
Perform a feasibility study on imagined acupuncture treatment of Chemotherapy-induced peripheral neuropathy (CIPN)

DETAILED DESCRIPTION:
We will perform a pilot study to assess the feasibility of Video-Guided Acupuncture Imagery Treatment (VGAIT) on CIPN symptoms in patients with stage I-III breast cancer with persistent CIPN after adjuvant chemotherapy. Participants will receive 16 sessions of VGAIT over 8 weeks remotely through the zoom. Study measures will be collected at the time of study enrollment, week 4, and week 8. The primary endpoints of the study will be 1) retention to treatment; 2) satisfaction for the intervention and 3) completion of study assessments.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* have histologically confirmed stage I-III breast cancer,
* have completed adjuvant taxane-based chemotherapy (alone or in combination), ,
* have an Eastern Cooperative Oncology Group performance status of 0 or 1, and reported grade 1 or greater CIPN symptoms for more than 2 weeks as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03.

Exclusion Criteria:

* concurrent chemotherapy (there were no limitations on time from the last paclitaxel administration),
* having metastatic or recurrent disease,
* history of preexisting peripheral neuropathy prior to chemotherapy,
* uncontrolled seizure disorder,
* unstable cardiac disease or myocardial infarction within 6 months prior to study entry, being pregnant or nursing, or having used acupuncture for CIPN within 6 months prior to study entry.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility related outcomes | 8 week
  Completion, satisfaction

SECONDARY OUTCOMES:
Patient Neurotoxicity Questionnaire (PNQ) | baseline, 8 week
  A tool designed to assess neurotoxic effects in patients who have undergone treatments such as chemotherapy
Functional Assessment of Cancer Therapy-Neurotoxicity subscale (FACT-NTX) | baseline, 8 week
  a widely used, validated instrument that assesses the impact of neuropathy on health-related quality of life
Brief Pain Inventory-short form (BPI-SF) | baseline, 8 week
  An instrument used to evaluate the severity of pain, including neuropathic pain, and the impact on the patient's daily functioning.
European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 (QLQ-C30) instrument | baseline, 8 week
  an instrument developed to assess the quality of life in cancer patients
MGH Acupuncture Sensation Scale (MASS) | after each intervention
  scale includes 12 descriptors of sensations frequently described during acupuncture treatment
Pain Catastrophizing Scale (PCS) | baseline, 8 week
  a 13-item self-report scale which measures pain-related rumination, magnification, and helplessness

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States